CLINICAL TRIAL: NCT06814691
Title: Evaluation of Analytical Thinking Skills and Reaction Tests of Female Football Players on Performance: Effects on In-Game Decision Making Processes
Brief Title: Effects on In-Game Decision Making Processes
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: E-85646034-604.01-93402
Record Dates: First submitted 2024-12-21; First posted 2025-02-07 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Athletic Injuries
Keywords: exercise
MeSH Terms: conditions — Athletic Injuries; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- football player: football player

SUMMARY:
This study aims to investigate the effects of analytical thinking skills and reaction speed on performance in female football players.

DETAILED DESCRIPTION:
This study aims to investigate the effects of analytical thinking skills and reaction speed on performance in female football players.

ELIGIBILITY:
Inclusion Criteria:

* Accepting the voluntary basis
* To be between the ages of 18-35
* To take part in professional football clubs
* Not having suffered any serious injury in the last 6 months
* To be able to participate in the Tampa Kinesiophobia Scale
* To be able to actively participate in technology-based tests such as decision-making simulations and Blazepod

Exclusion Criteria:

* Not accepting the voluntary basis
* Individuals who have had a surgical procedure in the last six months
* Use of NSAIDs and similar disease modifying drugs in the last month (Diaserein, Glucosamine etc.)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: The footballers who will take part in the study will be selected from players between the ages of 18-30, who are actively playing in professional football teams and have at least two years of experience.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Assessment of Analytical Thinking and Decision-Making Processes | day 1
  Female football players' analytical thinking skills will be evaluated through decision-making simulations and video-based training (VBT).
Assessment of Analytical Thinking and Decision-Making Processes-Accuracy | day 1
  Female football players' analytical thinking skills will be evaluated through decision-making simulations and video-based training (VBT).
Assessment of Analytical Thinking and Decision-Making Processes-Error Rates | day 1
  Female football players' analytical thinking skills will be evaluated through decision-making simulations and video-based training (VBT).
Tampa Scale of Kinesiophobia-Reaction Times | day 1
  The Tampa Scale of Kinesiophobia is a 17-item scale developed to assess fear of movement and reinjury. It includes parameters related to work activities, injury/reinjury, and fear-avoidance behaviors. The scale uses a 4-point Likert scoring system (1 = Strongly Disagree, 4 = Strongly Agree). After reversing the scores of items 4, 8, 12, and 16, a total score is calculated, ranging from 17 to 68, where higher scores indicate greater kinesiophobia.
Reaction Time Measurement (Using Blazepod) | day 1
  Blazepod devices will be used to measure the reaction speed and agility of female football players. Pods will be randomly placed and programmed to flash at specific intervals. Participants will be required to respond quickly to the flashing pods, with their reaction times recorded in milliseconds. Statistical data such as correct and incorrect response rates will also be obtained.
Y-Balance Test | day 1
  Evaluates balance by measuring reach distances in anterior, posteromedial, and posterolateral directions.
Push-Up Test | day 1
  Assesses upper body strength and endurance based on the number of push-ups performed.
Seated Ball Throw Test | day 1
  Measures upper body power by recording the distance a seated participant can throw a ball.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahçehir University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No